CLINICAL TRIAL: NCT00608634
Title: Phase 2a Randomized, Placebo-Controlled, Double-Blind Trial of Topical Perillyl Alcohol in Sun Damaged Skin
Brief Title: Topical Perillyl Alcohol in Treating Patients With Sun Damaged Skin and Actinic Keratoses
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Arizona Disease Control Research Commission (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CDR0000582634; P01CA027502 (NIH); P30CA023074 (NIH); UARIZ-HSC-04-27 (Other: UA IRB no.); UARIZ-POH-002 (Other: NCI)
Record Dates: First submitted 2008-02-05; First posted 2008-02-06 (Estimated); Results first posted 2015-04-01 (Estimated); Last update posted 2015-04-01 (Estimated); Status verified 2014-03

CONDITIONS: Precancerous Condition
Keywords: actinic keratosis
MeSH Terms: conditions — Precancerous Conditions; Keratosis, Actinic | interventions — perillyl alcohol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Patients apply a placebo cream topically to each dorsal forearm twice daily for 3 months in the absence of unacceptable toxicity.
  Interventions: Other: placebo
- Low Dose POH 0.30% (Experimental): Patients apply perillyl alcohol (POH) cream (0.3%) topically to each dorsal forearm twice daily for 3 months in the absence of unacceptable toxicity.
  Interventions: Drug: perillyl alcohol
- High Dose POH 0.76% (Experimental): Patients apply perillyl alcohol (POH) cream (0.76%) topically to each dorsal forearm twice daily for 3 months in the absence of unacceptable toxicity.
  Interventions: Drug: perillyl alcohol

INTERVENTIONS:
Drug: perillyl alcohol — Applied as topical cream
  Arms: High Dose POH 0.76%; Low Dose POH 0.30%
Other: placebo — Applied as topical cream
  Arms: Placebo

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as perillyl alcohol, work in different ways to stop the growth of abnormal cells, either by killing the cells or by stopping them from dividing. It is not yet known which dose of topical perillyl alcohol is more effective in stopping the development of cancer in sun damaged skin.

PURPOSE: This randomized phase II trial is studying high-dose topical perillyl alcohol to see how well it works compared with low-dose topical perillyl alcohol in treating patients with sun damaged skin and actinic keratoses.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To determine if topical administration of perillyl alcohol (POH) cream can reverse actinic damage as evidenced by normalization of quantitative skin histopathology scores in skin tissue biopsy samples from patients with moderate to severe sun damage.

Secondary

* To determine if topical POH can be administered safely to the forearms of these patients.

OUTLINE: Patients are randomized to 1 of 3 arms.

* Placebo: Patients apply a placebo cream topically to each dorsal forearm twice daily for 3 months in the absence of unacceptable toxicity.
* Low Dose: Patients apply perillyl alcohol (POH) cream (0.3%) topically to each dorsal forearm twice daily for 3 months in the absence of unacceptable toxicity.
* High Dose: Patients apply POH cream (0.76%) as in arm II. Patients undergo tissue sampling of the right or left dorsal forearm and of physician-selected representative actinic keratoses (AK) at baseline and after completion of study therapy. Tissue samples are assessed for changes in patterns of biomarker expression (i.e., p53, apoptosis, c-Fos histopathology) and karyometry. After completion of study therapy, patients undergo tissue sampling of the opposite forearm as well as blood sample collection to determine perillyl alcohol (POH) levels in blood and biopsy samples. Urine is also collected and analyzed for safety at the end of treatment. Digital photographs of the forearms and hands are obtained at baseline and after 3 months of study treatment. Optical coherence tomography imaging is also performed on pre- and post-biopsy sites to quantify the effect of POH on sun damage and AK in skin.

After completion of study treatment, patients are followed monthly.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Resident of Pima or adjoining Southern Arizona county

  * Patients outside of Pima County are also eligible
* Sun damaged skin as judged by the study physician and quantifiable, clinically diagnosed, and visible actinic keratoses (AK) on both dorsal forearms, with at least two AK on each arm

  * AK lesions must not be clustered, confluent, or too numerous to count accurately
  * Presence of AK on sites other than the test area allowed
* No significant inflammation or irritation of the skin of the upper extremities that is not clinically diagnosed as sun damage or AK
* Patients must agree to limit sun exposure as much as possible and may continue their normal pattern of sunscreen use

PATIENT CHARACTERISTICS:

Inclusion criteria:

* Females must not be of childbearing potential, and therefore must be post-menopausal or surgically sterile by hysterectomy
* Not pregnant or nursing

Exclusion criteria:

* Concurrent skin malignancy or disorder of the upper extremities

  * Patients with Squamous cell carcinoma or basal cell carcinoma in an area other than the test area are eligible upon excision of the Squamous cell carcinoma or basal cell carcinoma
* Patients who are immunosuppressed by virtue of medication or disease
* Serious concurrent illness that could interfere with study regimen
* Invasive cancer within the past 5 years

PRIOR CONCURRENT THERAPY:

* At least 30 days since prior topical medications to the skin of the upper extremities except for emollients or sunscreens
* At least 30 days since prior and no concurrent mega-doses of vitamins, defined as any of the following:

  * More than 5 times the recommended daily allowance
  * More than 5 capsules of multivitamins
  * 400 IU of vitamin E
  * 200 μg of selenium
  * 1 gm of vitamin C
* At least 6 months since prior and no concurrent therapy for squamous cell carcinoma (SCC) or basal cell carcinoma (BCC) anywhere in the test area (i.e., the forearms or hands)

  * Treatment for Squamous cell carcinoma or basal cell carcinoma on sites other than the test area is allowed
* At least 4 weeks since prior surgical biopsy, surgical excision, or cryotherapy for AK in the test area and the sites must have healed
* At least 6 months since prior topical treatment (e.g., 5-fluorouracil or imiquimod) for AK
* No concurrent therapy that may interfere with clinical evaluations
* No concurrent topical drug treatment (e.g., retinoids, aminolevulinic acid, diclofenac sodium, imiquimod, or fluorouracil) to any area of skin, including test area
* No concurrent enrollment in another clinical trial
* No concurrent topical citrus peel or consumption of citrus peel
* No chemotherapy for cancer within the past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2004-05; Primary Completion 2008-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Stratton, PhD, Study Chair — University of Arizona
Locations (1):
- Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Placbeo: Patients apply a placebo cream topically to each dorsal forearm twice daily for 3 months in the absence of unacceptable toxicity.
- High Dose POH 0.76%: Patients apply POH cream (0.76%) as in arm II.
Period: Overall Study
Arm/Group | Placbeo | Low Dose POH 0.30% | High Dose POH 0.76%
Started | 28 | 27 | 28
Completed | 26 | 26 | 27
Not Completed | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm I: Patients apply a placebo cream topically to each dorsal forearm twice daily for 3 months in the absence of unacceptable toxicity.
- Arm II: Patients apply perillyl alcohol (POH) cream (0.3%) topically to each dorsal forearm twice daily for 3 months in the absence of unacceptable toxicity.
- Arm III: Patients apply POH cream (0.76%) as in arm II.
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II | Arm III | Total
Number analyzed (Participants) | 28 | 27 | 28 | 83
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 14 | 10 | 13 | 37
  >=65 years | 14 | 17 | 15 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (9.9) | 68.8 (10.6) | 67.6 (10.9) | 67.7 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 5 | 20
  Male | 20 | 20 | 23 | 63
Region of Enrollment [Number; unit: participants]
  United States | 28 | 27 | 28 | 83

OUTCOME MEASURES:

1. Primary Outcome: Change in Histopathology Score of Sun Damaged Skin by Treatment Group
Description: The histopathologic scoring for skin biopsies from sun-damaged skin to assess the following seven characteristics: 1- atypia (levels 0, 1 & 2), 2- inflammation (grades 0, 1 & 2), 3- hyperkeratosis (loss of basket weave pattern of stratum corneum), 4- parakeratosis (present when there were >3 characteristic nuclei per 40:1 field in stratum corneum), 5- dyskeratosis (focal presence of cells with homogenous, pink cytoplasm n pyknotic nuclei), 6- epidermotropism (lymphocytes migration of >3 cells into epidermis, 7- loss of granular layer. All assessments were done using a 40:1 objective.
Time Frame: Baseline to 3 months
Population: change in histopathological scoring was calculated only for participants with baseline and end of study measurements. (n=79)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Low Dose POH 0.30% | High Dose POH 0.76%
Number analyzed (Participants) | 26 | 26 | 27
units on a scale | 0.4 (1.3) | -0.1 (1.3) | 0.1 (1.4)
Statistical Analysis 1: Comparison: Placebo vs Low Dose POH 0.30%; Test type: Superiority or Other; p = 0.10, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Placebo vs High Dose POH 0.76%; Test type: Superiority or Other; p = 0.41, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Skin Related Events From Perillyl Alcohol at Administered Doses by Participants
Description: The events do not have to be caused by the drug or therapy, and they may be mild, moderate, or severe. (NCI)
Time Frame: 3 months
Measure: Number; unit: participants
Groups:
- Low Dose 0.30% POH: Patients apply perillyl alcohol (POH) cream (0.3%) topically to each dorsal forearm twice daily for 3 months in the absence of unacceptable toxicity.
- High Dose 0.76% POH: Patients apply POH cream (0.76%) as in arm II.
Arm/Group | Placebo | Low Dose 0.30% POH | High Dose 0.76% POH
Number analyzed (Participants) | 28 | 27 | 28
participants
  No rash, redness, erythema | 16 | 12 | 13
  No flaking, crusting | 23 | 20 | 23
  No burning or stinging | 25 | 24 | 27
  No pruritus | 22 | 23 | 23
  Mild rash, redness, erythema | 11 | 14 | 15
  Mild flaking, crusting | 5 | 7 | 4
  Mild burning or stinging | 2 | 3 | 1
  Mild pruritus | 6 | 3 | 4
  Moderate rash, redness, erythema | 1 | 1 | 0
  Moderate flaking, crusting | 0 | 0 | 1
  Moderate burning or stinging | 1 | 0 | 0
  Moderate pruritus | 0 | 1 | 1
Statistical Analysis 1: Comparison: Placebo vs Low Dose 0.30% POH vs High Dose 0.76% POH; Test type: Superiority or Other; p > 0.05, Chi-squared

ADVERSE EVENTS:
Time Frame: 3 months for each participant.
Description: Standard Questionnaire
Groups:
- Low Dose POH 0.3%: Patients apply perillyl alcohol (POH) cream (0.3%) topically to each dorsal forearm twice daily for 3 months in the absence of unacceptable toxicity.
- High Dose POH 0.76%: Patients apply POH cream (0.76%) topically to each dorsal forearm twice daily for 3 months in the absence of unacceptable toxicity.
Arm/Group | Placebo | Low Dose POH 0.3% | High Dose POH 0.76%
Serious Adverse Events (participants affected / at risk) | 4/28 | 5/27 | 1/28
Other Adverse Events (participants affected / at risk) | 11/28 | 14/27 | 15/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=28) | Low Dose POH 0.3% (N=27) | High Dose POH 0.76% (N=28)
SCC in treatment area (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2) | 0 (0) — Biopsy sample clinically diagnosed as Actinic Keratoses (AKS), evaluated as squamous cell carcinoma in the histological evaluation.
SCC outside of treatment area (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) — One Squamous Cell Carcinoma on left ear (outside of treatment area). One Squamous Cell Carcinoma on cheek.
Stent Replacement (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) — Brief hospitalization for stent replacement
BCC outside of treatment area (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Basal Cell Carcinoma on cheek.
Bowel Obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Melanoma (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Not in test area
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=28) | Low Dose POH 0.3% (N=27) | High Dose POH 0.76% (N=28)
Mild Rash, Redness, Erythema (Skin and subcutaneous tissue disorders) | 11 (11) | 14 (14) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No